CLINICAL TRIAL: NCT05581238
Title: External Validation of the TRACK Allogeneic Transfusion Model in a Dutch Adult Cardiac Surgery Population, and the Effect on Discriminative Ability When Adding Anti-platelet Therapy
Brief Title: Validation of a Red Blood Cell Transfusion Prediction Model in a Low Transfusion Rate Population.
Acronym: TRACK-TCT
Status: Completed | Type: Observational
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, Renard Haumann, Principal Investigator, Medisch Spectrum Twente
Other Study IDs: Protocol_TRACK-TCT_v 2.0
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Platelet Aggregation; Blood Transfusion
Keywords: External validation; Blood transfusion; P2Y12 Receptor Inhibitor; Prediction Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TRACK: External validation of TRACK prediction model with 5 variables: age, weight, sex, pre-op HCT, Type of surgery.
- TRACK-TCT: New model development with 6 variables. 5 From the TRACK model: age, weight, sex, pre-op HCT, Type of surgery. A sixth variable will be added i.e.: pre-operative P2Y12 drug use
  Interventions: Other: TRACK-TCT

INTERVENTIONS:
Other: TRACK-TCT — An extra variable will be added to an existing prediction model. It is hypothesized that the predictive ability will improve and that better distinction could be made between patients with an increased risk for receiving blood transfusions.
  Groups: TRACK-TCT

SUMMARY:
The transfusion risk and clinical knowledge (TRACK) allogeneic blood transfusion prediction model was developed more than ten years ago and demonstrated good discriminative ability in patients with increased risk for allogeneic blood transfusion in an all Italian population. At the time of derivation, dual anti-platelet medication was suggested in the treatment of acute coronary syndrome, but not yet fully implemented.

The aim of this study is to externally validate the TRACK blood transfusion prediction model in the cardiac surgery population of Medisch Spectrum Twente Thoraxcentrum Twente. Additionally, the impact of adding the preoperative use of dual anti-platelet medication, as additional predictive factor, to the TRACK blood transfusion prediction model will be investigated.

DETAILED DESCRIPTION:
Cardiothoracic surgery is associated with increased perioperative blood loss and the need for allogeneic blood and blood product transfusions. This is due to three distinct factors, the invasive nature of the surgical procedures, the need for high dose anti-coagulation during extracorporeal circulation, and lastly the exposure of blood to the internal surface area of the heart-lung machine. Most cardiac patients use anti-platelet therapy before and after surgery, making hemostasis management in this specific patient population even more complex. European guidelines recommend administering anti-platelet therapy using Aspirin in combination with platelet receptor inhibitors such as Clopidogrel, Prasugrel or Ticagrelor, also known as dual anti-platelet therapy in patients with acute coronary syndrome.

Making distinct decisions regarding individual patient hemostasis management remains challenging. Decision making supported by prediction models, such as, EuroSCORE is well established in the cardiac surgery population. A few models pertaining specifically to allogeneic blood transfusion have been created and externally validated. Most of these prediction models perform reasonably well, predicting red blood cell transfusions with seventy-eighty percent accuracy, depending on the model and number of prediction factors used. Some are even excellent for predicting the chance of severe post-operative bleeding. As the transfusion of even one unit of allogeneic blood transfusion impacts mortality, the choice for the best feasible prediction model for routine clinical practice that reflects daily practice, uses a limited number of predictive factors, has a predictive capacity of more than seventy percent, and discriminates between risk groups for allogeneic blood transfusion is desirable.

Transfusion Risk and Clinical Knowledge (TRACK) model validation and optimization The TRACK model was developed more than ten years ago in an Italian adult cardiac surgery population. The decision to validate the TRACK model was based on its simplicity and relatively high predictive capacity, in comparison to other models with higher numbers of complex factors. This model has an allogeneic blood transfusion predictive capacity of seventy-two percent and uses a point system to divide patients into different risk groups, according to the total number of points allocated. During the derivation of this model, dual anti-platelet medication was included, but no significant association was found. In the twelve years since development, the popularity of dual anti-platelet medication used in acute coronary syndrome patients has significantly increased and its association with post-operative bleeding and allogeneic blood transfusion has been suggested.

Recent studies suggest that platelet activity may play a significant role in the prediction of post-operative bleeding, and one research group found that adding platelet activity to the CRUSADE score showed a significant increase in predicting risk of major bleeding in acute coronary syndrome patients. A re-evaluation of the association between dual anti-platelet (DAPT) and allogeneic blood transfusion is necessary. This will be done by the addition of DAPT as an extra predictive factor to the TRACK model, during external validation.

The negative association between mortality and transfusion products is well known. In addition, the related significant increase in hospital costs makes better perioperative hemostasis management crucial. Identifying cardiac surgery patients at risk for blood transfusion pre-operatively would aid clinicians in modifying the perioperative approach with goal the prevention of unnecessary allogeneic blood transfusion and the associated complications thereof.

Validating this model might aid clinicians in reducing allogeneic blood transfusions, transfusion complications and associated costs. Ultimately this might aid for development of patient specific transfusion strategies and new blood management protocols.

The aim of this study is to externally validate the TRACK blood transfusion prediction model in the cardiac surgery population of Medisch Spectrum Twente Thoraxcentrum Twente. Additionally, the impact of adding the preoperative use of dual anti-platelet medication will be studied, as additional predictive factor, to the TRACK blood transfusion prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving on-pump cardiac surgery

Exclusion Criteria:

* Patients who opted out for reuse of their data for scientific purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients, 18 years and older, who underwent any cardiac surgery with the use of a heart lung machine, between 1 January 2016 and 31 December 2021 in the Thoraxcentrum Twente, Medisch Spectrum Twente, Enschede.
Sampling Method: Non-Probability Sample
Enrollment: 6428 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
External validation TRACK blood prediction Model (TRACK) | 1 year
  Does adding P2Y12 inhibitors as extra variable to the TRACK model after validation improve the predictive capacity? This will be done by validation of the TRACK model in the cardiac surgery population of TCT by calculating the discriminative ability. The change in discriminative ability, after correction for optimism, when the pre-operative use of P2Y12 inhibitors is added as extra variable will be assessed and the net improvement in reclassification will be calculated.
Evaluation of the change in predictive capacity when adding P2Y12 as extra variable (TRACK-TCT) | 1 year
  Does adding P2Y12 inhibitors as extra variable to the TRACK model after validation improve the predictive capacity? This will be done by validation of the TRACK model in the cardiac surgery population of TCT by calculating the discriminative ability. The change in discriminative ability, after correction for optimism, when the pre-operative use of P2Y12 inhibitors is added as extra variable will be assessed and the net improvement in reclassification will be calculated.

SECONDARY OUTCOMES:
Male vs Female | 1 year
  How does the performance of the model change in an all-male and all-female population.
Post operative complication in patients that received a blood transfusion | 1 year
  Does allogeneic blood transfusion increase the risk of post-operative complications or thromboembolic events?
Mortality difference in patients that received a blood transfusion | 1 year
  What is the difference in 30-day mortality between patients receiving allogeneic blood transfusions and patients that does not?

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Halfwerk, MD PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Thoraxcentrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be made openly available in a repository according to FAIR (Findable, Accessible, Interoperable, Reproducible) guidelines.
Supporting Information: Analytic Code
Time Frame: During this year (2024)

REFERENCES:
- [Background] Gorlinger K, Shore-Lesserson L, Dirkmann D, Hanke AA, Rahe-Meyer N, Tanaka KA. Management of hemorrhage in cardiothoracic surgery. J Cardiothorac Vasc Anesth. 2013 Aug;27(4 Suppl):S20-34. doi: 10.1053/j.jvca.2013.05.014. PMID 23910533
- [Background] Raphael J, Mazer CD, Subramani S, Schroeder A, Abdalla M, Ferreira R, Roman PE, Patel N, Welsby I, Greilich PE, Harvey R, Ranucci M, Heller LB, Boer C, Wilkey A, Hill SE, Nuttall GA, Palvadi RR, Patel PA, Wilkey B, Gaitan B, Hill SS, Kwak J, Klick J, Bollen BA, Shore-Lesserson L, Abernathy J, Schwann N, Lau WT. Society of Cardiovascular Anesthesiologists Clinical Practice Improvement Advisory for Management of Perioperative Bleeding and Hemostasis in Cardiac Surgery Patients. Anesth Analg. 2019 Nov;129(5):1209-1221. doi: 10.1213/ANE.0000000000004355. PMID 31613811
- [Background] Task Force on Patient Blood Management for Adult Cardiac Surgery of the European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology (EACTA); Boer C, Meesters MI, Milojevic M, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Pagano D. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):88-120. doi: 10.1053/j.jvca.2017.06.026. Epub 2017 Sep 30. No abstract available. PMID 29029990
- [Background] Karkouti K, Wijeysundera DN, Yau TM, Beattie WS, Abdelnaem E, McCluskey SA, Ghannam M, Yeo E, Djaiani G, Karski J. The independent association of massive blood loss with mortality in cardiac surgery. Transfusion. 2004 Oct;44(10):1453-62. doi: 10.1111/j.1537-2995.2004.04144.x. PMID 15383018
- [Background] Ranucci M, Bozzetti G, Ditta A, Cotza M, Carboni G, Ballotta A. Surgical reexploration after cardiac operations: why a worse outcome? Ann Thorac Surg. 2008 Nov;86(5):1557-62. doi: 10.1016/j.athoracsur.2008.07.114. PMID 19049749
- [Background] Khan B, Islam MU, Ahmad I, Rehman MU. Modifiable Risk Factors associated with Post-Operative Bleeding and transfusion requirements in Cardiac Surgery. Pak J Med Sci. 2022 Mar-Apr;38(4Part-II):855-861. doi: 10.12669/pjms.38.4.5685. PMID 35634631
- [Derived] Haumann R, Plonek T, Niesten E, Maaskant J, Arens J, van der Palen J, Halfwerk F. Validation and optimization of a blood transfusion prediction model for low transfusion rate adult cardiac surgery. Perfusion. 2025 Apr 19:2676591251334903. doi: 10.1177/02676591251334903. Online ahead of print. PMID 40252042